CLINICAL TRIAL: NCT05561322
Title: Third Year Post-surgical Evaluation of Onset of Adjacent Segment Disc Degeneration in the Lumbar Spine According to the Initial Technique (Spinal Fusion Versus Lumbar Arthroplasty With Disc Replacement). A Monocentric Prospective Non-randomized Cohort Study.
Brief Title: 3rd-year Post-surgical Evaluation of Adjacent Segment Disc Degeneration Onset in Lumbar Spine (Spinal Fusion vs. Lumbar Arthroplasty With Disc Replacement)
Acronym: ARTHRO-DEGE
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2018-02/PK-01; RCB no. (Registry Identifier: 2019-A01035-52)
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Spine Surgery
Keywords: Arthroplasty; Arthrodesis; Disc degeneration; Lumbar spine; Spinal fusion
MeSH Terms: conditions — Ankylosis; Intervertebral Disc Degeneration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal fusion patients: Patients who have undergone spinal fusion surgery and have had at least 3 years of follow-up.
  Interventions: Other: Consultation involving pain evaluation, questionnaires and the Lasègue Manoeuver; Other: Magnetic Resonance Imaging of the lumbar spine
- Lumbar arthroplasty patients: Patients who have undergone lumbar arthroplasty with disc replacement and have had at least 3 years of follow-up.
  Interventions: Other: Consultation involving pain evaluation, questionnaires and the Lasègue Manoeuver; Other: Magnetic Resonance Imaging of the lumbar spine

INTERVENTIONS:
Other: Consultation involving pain evaluation, questionnaires and the Lasègue Manoeuver — Raising the lower limb with the knee in extension reproduces sciatica pain if there is an impression of discal pain with its origin at the roots of the sciatica nerve L5 and S1. This test is evaluated by the degree of elevation of the lower limb relative to the examination table. During the Lasègue manoeuvre the sciatica pain is improved during dorsal flexion of the foot.The doctor notes whether the Lasègue manoeuvre done on the healthy side exacerbates the pain on the opposite side. It is said that contralateral Lasègue sign is positive.
  Other Names: Lasègue manoeuver
Other: Magnetic Resonance Imaging of the lumbar spine — Sagittal proton density-weighted Dixon sequence on the lumbar spine and axial T2-weighted spin echo sequence on the lumbar discs.

SUMMARY:
The main objective of the study is to compare the onset of adjacent segment disk degeneration in two groups of patients (one "spinal fusion group" and one "lumbar arthroplasty with disc replacement" group) with each patient acting as their own control for either group under study and more than three years of follow-up.

DETAILED DESCRIPTION:
This is a non-randomized prospective monocentric open cohort study. Patients whose surgical intervention goes back to more than 3 years will be preselected from the KEOPS database and contacted by phone. Information on the study and its restrictions is delivered to the patient. The investigator organizes the inclusion visit. The patient is seen for consultation by the orthopedic surgeon (inclusion visit /end of research) ; the information notice is given to the patient who is free to ask questions about the study. The patient's consent is collected. The investigator proceeds with a clinical examination (the Lasègue manoeuver), evaluates pain (EVN, DN4) and administers four different questionnaires .

The patient is then oriented towards the imaging department where he/she will have the benefit of and Magnetic Resonance Imaging and also a spinal X-ray(front and profile ; Roussouly classification).

The patient's participation in the study ends once the examination is over. The consultation in the orthopedic department and the imaging session will be planned in such a way that they can be performed all on the same day.

The study program provides for 12 months of inclusion and 4 months of data management, statistical analysis and writing up the report on the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have given written, informed consent.
* All patients covered by a health insurance scheme.
* All patients aged over 18.
* All patients operated with a lumbar spine disk prosthesis or vertebral arthrodesis with an anterior approach at the Orthopedic, Traumatology and Spine Surgery Department of Nimes University Hospital, France, at least 3 years previously.
* All patients who have undergone initial MRI before surgery.

Exclusion Criteria:

* Any patient taking part in a category 1 interventional study and in an exclusion period determined by a previous study.
* Any patient under legal protection, guardianship or tutorship.
* Any patient who refuses to sign the consent form.
* Any patient for whom it is impossible to give clear information.
* Any patient with contra-indications for Magnetic Resonance Imaging such as an incompatible pacemaker, claustrophobia, metal apparatus or prosthetic hip.
* Any patient with a septic complication.
* Any patient with instrumentation or posterior arthrodesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients being managed by the Orthopedic,Traumatology and Spine Surgery Department of Nimes University Hospital, France, taken from the hospital's KEOPS database. Patients in the study have all undergone lumbar disk surgery with either a prosthetic disk or arthrodesis with an anterior approach and have at least 3 years of follow-up.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of adjacent segment disc degeneration in spinal fusion patients | Day of consultation, at least 3 years after the initial surgery
  The onset of adjacent segment disc degeneration in spinal fusion patients will be evaluated with magnetic resonance imaging.
Evaluation of adjacent segment disc degeneration in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  Adjacent segment disc degeneration in lumbar arthroplasty patients will be evaluated with magnetic resonance imaging.

SECONDARY OUTCOMES:
Adjacent disc degeneration in spinal fusion patients according to the MODIC classification | Day of consultation, at least 3 years after surgery
  The classification by Michael MODIC evaluates the stage of disk degeneration seen with magnetic resonance imaging as follows :
  Stage 0 : Disc appears black on sequences 1 and 2. Dehydration of disk without retraction of the vertebral end plates.
  Stage 1 : Disc appears black on sequence 1 but white on sequence 2. Inflammatory reaction on vertebral end plates. Swollen aspect.
  Stage 2: Disc appears white on both sequences 1 and 2. Fatty reaction of vertebral end plates. Fatty aspect.
  Stage 3: Disc appears black on both sequences 1 and 2. Bony sclerosis.
Adjacent disk degeneration in lumbar arthroplasty patients according to the MODIC classification | Day of consultation, at least 3 years after surgery
  The classification by Michael MODIC evaluates the stage of disc degeneration seen with magnetic resonance imaging as follows :
  Stage 0 : Disc appears black on sequences 1 and 2. Dehydration of disc without retraction of the vertebral end plates.
  Stage 1 : Disc appears black on sequence 1 but white on sequence 2. Inflammatory reaction on vertebral end plates. Swollen aspect.
  Stage 2: Disc appears white on both sequences 1 and 2. Fatty reaction of vertebral end plates. Fatty aspect.
  Stage 3: Disc appears black on both sequences 1 and 2. Bony sclerosis.
Quantification of the evolution of adjacent disk degeneration in spinal fusion patients according to the modified Pfirmann classification. | Day of consultation, at least 3 years after surgery
  The modified Pfirmann classification is used to grade disc degeneration as seen on magnetic resonance imaging with T2-weighted sagittal or STIR sequences. Grade 1 corresponds to a healthy disc rarely observed in adults. Grade 5 corresponds to disk collapse.
Quantification of the evolution of adjacent disk degeneration in lumbar arthroplasty patients according to the modified Pfirmann classification. | Day of consultation, at least 3 years after surgery
  The modified Pfirmann classification is used to grade disc degeneration as seen on magnetic resonance imaging with T2-weighted sagittal or STIR sequences. Grade 1 corresponds to a healthy disc rarely observed in adults. Grade 5 corresponds to disk collapse.
Disc degeneration count per spinal fusion patient | Day of consultation, at least 3 years after surgery
  The number of points of degeneration, just above or just below the operated segment, will be counted for each patient.
Disc degeneration count per lumbar arthroplasty patient | Day of consultation, at least 3 years after surgery
  The number of points of degeneration, just above or just below the operated segment, will be counted for each patient.
Weishaupt classification of disc degeneration in spinal fusion patients | Day of consultation, at least 3 years after surgery
  The Weishaupt classification classifies arthritis of the lumbar facet joints as follows:
  Grade 0: Normal facet joint space (2±4 mm width) Grade 1: Narrowing of the facet joint space (< 2 mm) and/or small osteophytes and/or mild hypertrophy of the articular process Grade 2: Narrowing of the facet joint space and/or moderate osteophytes and/or moderate hypertrophy of the articular process and/or mild subarticular bone erosions Grade 3: Narrowing of the facet joint space and/or large osteophytes and/or severe hypertrophy of the articular process and/or severe subarticular bone erosions and/or subchondral cysts
Weishaupt classification of disc degeneration in lumbar arthroplasty patients patients | Day of consultation, at least 3 years after surgery
  The Weishaupt classification classifies arthritis of the lumbar facet joints as follows:
  Grade 0: Normal facet joint space (2±4 mm width) Grade 1: Narrowing of the facet joint space (< 2 mm) and/or small osteophytes and/or mild hypertrophy of the articular process Grade 2: Narrowing of the facet joint space and/or moderate osteophytes and/or moderate hypertrophy of the articular process and/or mild subarticular bone erosions Grade 3: Narrowing of the facet joint space and/or large osteophytes and/or severe hypertrophy of the articular process and/or severe subarticular bone erosions and/or subchondral cysts
Hadar classification in spinal fusion patients | Day of consultation, at least 3 years after surgery
  Backache has an effect on the muscles provoking a gradual degeneration of muscle fat. Hadar proposes a 3-stage scale to classify the fibroadipose tissue.
Hadar classification in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  Backache has an effect on the muscles provoking a gradual degeneration of muscle fat. Hadar proposes a 3-stage scale to classify the fibroadipose tissue
Re-intervention rate among spinal fusion patients | Day of consultation, at least 3 years after surgery
  The number of re-interventions among spinal fusion patients will be recorded as a percentage.
Re-intervention rate among lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  The number of re-interventions among lumbar arthroplasty patients will be recorded as a percentage.
Evolution of pain among spinal fusion patients | Day of consultation, at least 3 years after surgery
  The DN4 hetero-questionnaire (" Neuropathic pain in 4 Questions ") is validated in French and evaluates the possible presence of neuropathic-type pain in a patient (Bouhassira et al. 2005). It consists of 4 questions (2 at the interview, 2 during the examination and 10 items for which the patient has to answer YES or NO. Each " YES" validates one point, each " NO " does not validate a point. If the score is ≥4,the test is positive.
Evolution of pain among lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  The DN4 hetero-questionnaire (" Neuropathic pain in 4 Questions ") is validated in French and evaluates the possible presence of neuropathic-type pain in a patient (Bouhassira et al. 2005). It consists of 4 questions (2 at the interview, 2 during the examination and 10 items for which the patient has to answer YES or NO. Each " YES" validates one point, each " NO " does not validate a point. If the score is ≥4,the test is positive.
Percentage incapacity according to the Oswestry Disability Index in spinal fusion patients. | Day of consultation, at least 3 years after surgery
  The Oswestry Disability Index is one of the most widely-used disability scales in the Anglophone world used to evaluate functional incapacity in patients with backache. It may be used not only in clinical studies but also by the General Practitioner to evaluate the evolution of a patient's functional incapacity. It contains 10 sections and at least 8 must be completed in order for the score to be calculable. It is expressed as percentage incapacity by multiplying by two the sum of the answers graduated 0 to 5 for each item. It has been validated in English ( Fisher & Johnston 1997; Little et MacDonald 1994; Fritz et Irrgang 2001; Grönblad et al. 1993; Fairbank and Pynsent 2000) and its French translation was validated in 2008 (Vogler et al. 2008).
Percentage incapacity according to the Oswestry Disability Index in lumbar arthroplasty patients. | Day of consultation, at least 3 years after surgery
  The Oswestry Disability Index is one of the most widely-used disability scales in the Anglophone world used to evaluate functional incapacity in patients with backache. It may be used not only in clinical studies but also by the General Practitioner to evaluate the evolution of a patient's functional incapacity. It contains 10 sections and at least 8 must be completed in order for the score to be calculable. It is expressed as percentage incapacity by multiplying by two the sum of the answers graduated 0 to 5 for each item. It has been validated in English ( Fisher & Johnston 1997; Little et MacDonald 1994; Fritz et Irrgang 2001; Grönblad et al. 1993; Fairbank and Pynsent 2000) and its French translation was validated in 2008 (Vogler et al. 2008).
Fears and Avoidance Beliefs Questionnaire in spinal fusion patients | Day of consultation, at least 3 years after surgery
  The notions of apprehension-avoidance of beliefs font part of the psychosocial factors associated with the onset, maintenance and reinforcement of the chronic pain process. Their evaluation is made with the FABQ questionnaire whose original English version was validated in 1993 by Waddell et al. (1993) and the French version in 2004 (Chaory et al.2004). The patient's fears, beliefs and avoidance attitudes are predictive of the result and observance of treatment, particularly functional restoration programs (Pfingsten et al. 2000). The FABQ is a self-questionnaire with 16 items rated 0 to 6 on a Likert scale (0 = absolutely disagree, 6 = completely agree) ; the questions focus on the appreciation of notions of apprehension relative to professional activities and other physical activities. It takes about 10 minutes to complete the questionnaire. A high score represents a high rate of fears and beliefs.
Fears and Avoidance Beliefs Questionnaire in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  The notions of apprehension-avoidance of beliefs font part of the psychosocial factors associated with the onset, maintenance and reinforcement of the chronic pain process. Their evaluation is made with the FABQ questionnaire whose original English version was validated in 1993 by Waddell et al. (1993) and the French version in 2004 (Chaory et al.2004). The patient's fears, beliefs and avoidance attitudes are predictive of the result and observance of treatment, particularly functional restoration programs (Pfingsten et al. 2000). The FABQ is a self-questionnaire with 16 items rated 0 to 6 on a Likert scale (0 = absolutely disagree, 6 = completely agree) ; the questions focus on the appreciation of notions of apprehension relative to professional activities and other physical activities. It takes about 10 minutes to complete the questionnaire. A high score represents a high rate of fears and beliefs.
Lasègue manoeuvre in spinal fusion patients | Day of consultation, at least 3 years after surgery
  This provocation test is very specific to radicular sciatica . Raising the lower limb with the knee in extension, reproduces sciatica pain if there is an impression of disk pain with its origin at the roots of the sciatica nerve L5 and S1. This test is evaluated by the degree of elevation of the lower limb relative to the examination table. During the Lasègue manoeuvre the sciatica pain is improved during dorsal flexion of the foot.The doctor notes whether the Lasègue manoeuvre done on the healthy side exacerbates the pain on the opposite side. It is said that contralateral Lasègue sign is positive.
Lasègue manoeuvre in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  This provocation test is very specific to radicular sciatica . Raising the lower limb with the knee in extension, reproduces sciatica pain if there is an impression of disk pain with its origin at the roots of the sciatica nerve L5 and S1. This test is evaluated by the degree of elevation of the lower limb relative to the examination table. During the Lasègue manoeuvre the sciatica pain is improved during dorsal flexion of the foot.The doctor notes whether the Lasègue manoeuvre done on the healthy side exacerbates the pain on the opposite side. It is said that contralateral Lasègue sign is positive.
Results of the SF-12 Quality of Life questionnaire in spinal fusion patients | Day of consultation, at least 3 years after surgery
  This quality of life self-evaluation scale is a short version of the SF-36 and gives two scores: one mental and social quality of life score, and one physical quality of life score (Ware et al. 1996). For the scoring (1) each answer to 12 items must be converted into standardized values both for the mental and social score and for the physical score, (2) the 12 standardized values obtained for the mental et social score are added together and (3) 60,75781 is added on to get the mental et social quality of life score. Then, the 12 standardized values obtained for the physical score are added together and 56,57706 is added on to get the physical quality of life score.
Results of the SF-12 Quality of Life questionnaire in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  This quality of life self-evaluation scale is a short version of the SF-36 and gives two scores: one mental and social quality of life score, and one physical quality of life score (Ware et al. 1996). For the scoring (1) each answer to 12 items must be converted into standardized values both for the mental and social score and for the physical score, (2) the 12 standardized values obtained for the mental et social score are added together and (3) 60,75781 is added on to get the mental et social quality of life score. Then, the 12 standardized values obtained for the physical score are added together and 56,57706 is added on to get the physical quality of life score.
Results of the Patient Global Impression of Change scale in spinal fusion patients | Day of consultation, at least 3 years after surgery
  The Patient Global Impression of Change scale is a self-questionnaire on satisfaction regarding the change brought by the treatment to daily activities, symptoms and quality of life in relation to chronic pain. This scale has been validated in French (Le Gal et al. 2010) and consists of 7 points. The patients are classified into 3 categories according to their score (Rampakakis et al. 2015): deterioration (a score of 1 to 3), stable (score of 4), improvement (score of 5 to 7).
Results of the Patient Global Impression of Change scale in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  The Patient Global Impression of Change scale is a self-questionnaire on satisfaction regarding the change brought by the treatment to daily activities, symptoms and quality of life in relation to chronic pain. This scale has been validated in French (Le Gal et al. 2010) and consists of 7 points. The patients are classified into 3 categories according to their score (Rampakakis et al. 2015): deterioration (a score of 1 to 3), stable (score of 4), improvement (score of 5 to 7).
MRI data acquisition in spinal fusion patients | Day of consultation, at least 3 years after surgery
  A 3T MRI scanner (Magnetom Skyra, Siemens Healthcare) equipped with a 32-channel head coil will be used to obtain the following sequences: sagittal proton density-weighted Dixon sequencing on the lumbar spine and axial T2-weighted spin echo sequencing on the lumbar discs.
MRI data acquisition in lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  A 3T MRI scanner (Magnetom Skyra, Siemens Healthcare) equipped with a 32-channel head coil will be used to obtain the following sequences: sagittal proton density-weighted Dixon sequencing on the lumbar spine and axial T2-weighted spin echo sequencing on the lumbar discs.
Body Mass Index of spinal fusion patients | Day of consultation, at least 3 years after surgery
  The patient's weight and height will be noted in an observation booklet and the patient's body mass index will be calculated via a computer (in kg/m2)
Body Mass Index of lumbar arthroplasty patients | Day of consultation, at least 3 years after surgery
  The patient's weight and height will be noted in an observation booklet and the patient's body mass index will be calculated via a computer (in kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France